CLINICAL TRIAL: NCT02819323
Title: A Safety and Efficacy Study of a Bowel Cleansing Preparation (BLI800) in Pediatric Subjects Undergoing Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BLI800-502
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- BLI800 high dose (Experimental): BLI800 bowel preparation (high dose)
  Interventions: Drug: BLI800
- BLI800 low dose (Experimental): BLI800 bowel preparation (low dose)
  Interventions: Drug: BLI800
- PEG-ELS (Active Comparator): PEG based bowel preparation
  Interventions: Drug: PEG-ELS

INTERVENTIONS:
Drug: PEG-ELS — polyethylene glycol based bowel preparation
  Arms: PEG-ELS
Drug: BLI800 — BLI800 bowel preparation
  Arms: BLI800 high dose; BLI800 low dose

SUMMARY:
The objective of this study is to compare the safety, tolerance and efficacy of BLI800 to a PEG based preparation prior to colonoscopy in adolescent patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 12 to 16 (inclusive)
2. Undergoing colonoscopy for routinely accepted indications, including (but not limited to):

   * Subjected inflammatory bowel disease (IBD) or IBD follow-up
   * Lower gastrointestinal bleeding
   * Suspected colitis (allergic or other)
   * Abdominal pain
   * Chronic diarrhea
   * Cancer surveillance
   * Anemia of unknown etiology
   * Abnormal endosonography or manometry
   * Evaluation of barium enema results
3. If female, and of child-bearing potential, subject must use an acceptable form of birth control or remain abstinent for the duration of the study.
4. Negative pregnancy test at screening, if applicable
5. In the Investigator's judgment, caregiver is mentally competent to provide informed consent for their child to participate in the study.

Exclusion Criteria:

1. Subjects with known or suspected ileus, impaction, severe ulcerative colitis, acute peritonitis, gastrointestinal obstruction, gastric retention (gastroparesis), bowel perforation, toxic colitis or megacolon.
2. Subjects who had previous significant gastrointestinal surgeries.
3. Subjects with increased risk of bowel perforation, including connective tissue disorders, toxic dilation of the bowel or recent bowel surgery.
4. Subjects with uncontrolled pre-existing electrolyte abnormalities, or those with clinically significant electrolyte abnormalities based on Visit 1 laboratory results, such as hypernatremia, hyponatremia, hyperphosphatemia, hypokalemia, hypocalcemia, uncorrected dehydration, or those secondary to the use of diuretics or angiotensin converting enzyme (ACE) inhibitors.
5. Subjects with bleeding disorders and/or impaired platelet function, or neutropenia.
6. Subjects with a prior history of renal, liver or cardiac insufficiency (including congestive heart failure or other significant cardiac abnormality)
7. Subjects with estimated glomerular filtration rate (GFR) below normal range (less than 70 ml/min/1.73m2)
8. Subjects required to take any other oral medication within 3 hours of dosing until completion of both doses.
9. Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
10. Subjects with tendency for nausea and/or vomiting, or that have known swallowing disorders.
11. Subjects for whom intake of substances is likely to affect gastrointestinal motility or urinary flow rate.
12. Subjects undergoing colonoscopy for foreign body removal and/or decompression.
13. Subjects with an abnormal ECG result at Visit 1.
14. Subjects who are pregnant or lactating, or intending to become pregnant during the study.
15. Subjects of childbearing potential who refuse a pregnancy test.
16. Subjects with a history of hypersensitivity to any preparation components.
17. Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures and history of major medical/psychiatric conditions that would compromise the safety of the study.
18. Subjects who have participated in an investigational surgical, drug, or device study within the past 30 days.
19. Subjects who withdraw consent before completion of Visit 1 procedures.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2016-06; Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, Study Director — Braintree Laboratories, Inc.
Locations (27):
- United States (27):
  - Braintree Research Site 27, Mobile, Alabama
  - Braintree Research Site 30, Tucson, Arizona
  - Braintree Research Site 23, Orange, California
  - Braintree Research Site 16, San Francisco, California
  - Braintree Research Site 5, Gainesville, Florida
  - Braintree Research Site 24, Jacksonville, Florida
  - Braintree Research Site 21, Orlando, Florida
  - Braintree Research Site 2, Atlanta, Georgia
  - Braintree Research Site 13, Chicago, Illinois
  - Braintree Research Site 3, Park Ridge, Illinois
  - Braintree Research Site 26, Indianapolis, Indiana
  - Braintree Research Site 25, Minneapolis, Minnesota
  - Braintree Research Site 18, Rochester, Minnesota
  - Braintree Research Site 1, Flowood, Mississippi
  - Braintree Research Site 9, Buffalo, New York
  - Braintree Research Site 28, New York, New York
  - Braintree Research Site 19, New York, New York
  - Braintree Research Site 32, The Bronx, New York
  - Braintree Research Site 6, Pittsburgh, Pennsylvania
  - Braintree Research Site 20, Memphis, Tennessee
  - Braintree Research Site 34, Plano, Texas
  - Braintree Research Site 22, Salt Lake City, Utah
  - Braintree Research Site 10, Burlington, Vermont
  - Braintree Research Site 17, Norfolk, Virginia
  - Braintree Research Site 4, Roanoke, Virginia
  - Braintree Research Site 11, Seattle, Washington
  - Braintree Research Site 14, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BLI800 High Dose: BLI800 bowel preparation (high dose)
  BLI800: BLI800 bowel preparation (6 oz)
- BLI800 Low Dose: BLI800 bowel preparation (low dose)
  BLI800: BLI800 bowel preparation (4.5 oz)
Period: Overall Study
Arm/Group | BLI800 High Dose | BLI800 Low Dose | PEG-ELS
Started (Safety population - all subjects that took preparation.) | 31 | 28 | 32
Completed | 26 | 26 | 31
Not Completed | 5 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety population - all subjects that took preparation.
Groups:
- Total: Total of all reporting groups
Arm/Group | BLI800 High Dose | BLI800 Low Dose | PEG-ELS | Total
Number analyzed (Participants) | 31 | 28 | 32 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.2) | 14.5 (1.4) | 14.4 (1.4) | 14.5 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 15 | 52
  Male | 12 | 10 | 17 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 3 | 9
  Not Hispanic or Latino | 27 | 26 | 29 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 9 | 15
  White | 27 | 24 | 20 | 71
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 31 | 28 | 32 | 91

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Subjects With Successful Bowel Cleansing
Description: Cleansing is rated by a blinded colonoscopist on a 4 point scale (1=poor to 4 = excellent)
Time Frame: 2 days
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | BLI800 High Dose | BLI800 Low Dose | PEG-ELS
Number analyzed (Participants) | 31 | 27 | 32
Participants | 25 | 22 | 19
Statistical Analysis 1: Comparison: BLI800 Low Dose vs PEG-ELS; Test type: Non-Inferiority — Non-inferiority margin = 10%; p = 0.003, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: BLI800 High Dose vs PEG-ELS; Test type: Non-Inferiority — Non-inferiority margin = 10%; p = 0.003, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: BLI800 Low Dose vs PEG-ELS; Test type: Superiority; p = 0.046, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: BLI800 High Dose vs PEG-ELS; Test type: Superiority; p = 0.089, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 30 days
Description: Patients were directly queried for the expected bowel preparation symptoms of abdominal distension, abdominal pain, nausea and vomiting.
Arm/Group | BLI800 High Dose | BLI800 Low Dose | PEG-ELS
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/28 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/28 | 1/32
Other Adverse Events (participants affected / at risk) | 29/31 | 26/28 | 29/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI800 High Dose (N=31) | BLI800 Low Dose (N=28) | PEG-ELS (N=32)
alcohol intoxication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Accidental Tylenol Ingestion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLI800 High Dose (N=31) | BLI800 Low Dose (N=28) | PEG-ELS (N=32)
Abdominal distension (Gastrointestinal disorders) | 20 (20) | 9 (9) | 17 (17)
Abdominal pain upper (Gastrointestinal disorders) | 17 (17) | 16 (16) | 20 (20)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 23 (23) | 16 (16) | 27 (27)
Vomiting (Gastrointestinal disorders) | 6 (6) | 8 (8) | 12 (12)
Headache (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Anion gap increased (Investigations) | 3 (3) | 3 (3) | 2 (2)
Bacterial test positive (Investigations) | 2 (2) | 2 (2) | 0 (0)
Blood bicarbonate decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 2 (2) | 1 (1) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Anion gap decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT02819323/Prot_SAP_000.pdf